CLINICAL TRIAL: NCT04969536
Title: Metabolomic Impacts of Branched-chain Amino Acid Supplementation During Endurance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: M.J. Murdoch Charitable Trust (Unknown); Kreighbaum Endowment (Unknown)
Responsible Party: Principal Investigator, Mary Miles, Professor, Montana State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: DF081319
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Branch-chained amino acids; Endurance exercise; Metabolomics; Serotonin
MeSH Terms: interventions — Amino Acids

STUDY DESIGN:
Intervention Model Description: 60 minutes of moderate (65% of VO2max) endurance exercise with either a branched chain amino acid supplement or a placebo consumed immediately prior to and 30 minutes into the exercise bout.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Branched chain amino acid supplementation (Experimental): Consumption of 8 ounces of water with addition of 2.5 g of leucine, 1.25 g of isoleucine, and 1.25 g of valine immediately prior to and again 30 minutes into a 60 minute treadmill run at 65% of VO2max.
  Interventions: Dietary Supplement: Branched Chain Amino Acids
- Placebo (Placebo Comparator): Consumption of 8 ounces of a flavor matched beverage sweetened with a sucralose-based drink mix immediately prior to and again 30 minutes into a 60 minute treadmill run at 65% of VO2max.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Branched Chain Amino Acids — Supplementation with 8 g Nutrex Research Amino Acid Drive BCAA in 8 ounces of water once each immediately pre-exercise and after 30 minutes of exercise
  Arms: Branched chain amino acid supplementation
Other: Placebo — Supplementation with 2.0 milliliters of a sucralose-based drink mix with 8 ounces of water once each immediately pre-exercise and after 30 minutes of exercise
  Arms: Placebo

SUMMARY:
The overall goal of this investigation was to determine the impact of branch-chained amino acids (BCAAs) supplementation on serotonin and associated metabolites during endurance exercise on healthy individuals. Specifically, despite the strong theoretical basis for supplementation of BCAAs to attenuate serotonin production and fatigue during exercise, most human clinical trials have failed to demonstrate these benefits. To shed light on this discrepancy, the purpose of this study was to measure the impact of BCAA supplementation on serotonin and associated metabolites during exercise.

To achieve this purpose, investigators determined the effects of the consumption of a BCAA beverage on endurance exercise performance and serum metabolites. The supplementation protocol consisted of two trials in which each participant consumed 8 grams of BCAA supplement in a beverage or a placebo in randomized order. It was hypothesized that post-exercise metabolites would differ between BCAA and placebo conditions.

DETAILED DESCRIPTION:
Research Design This study utilized a randomized, placebo-controlled, double-blind crossover design comparing supplementation of BCAA versus placebo beverages consumed immediately before and halfway through a 60-minute run at 65% of maximal aerobic capacity. To isolate the impact of BCAA on serotonin and metabolism during exercise, blood samples were collected immediately before and after exercise. A targeted metabolomic analysis was designed for BCAA to verify supplementation induced increases in serum concentration, as well as for serotonin to assess impacts of BCAAs. Untargeted metabolomic analysis was performed to identify global metabolic impacts of BCAA supplementation on metabolism during endurance exercise.

Maximal Aerobic Capacity A graded exercise test was used to measure maximal oxygen consumption (VO2max) using a motorized treadmill. Each participant was fitted with an electronic heart rate (HR) monitor, a mouthpiece and a two-way non-rebreathing tube and a nose clip, all of which were attached to a standard laboratory metabolic cart (TrueOne 2400, ParvoMedics, Sandy, Utah). Participants self-selected a speed between 5 and 7.5 mph and began running at a 0% incline. Each minute, the treadmill incline was increased by 1.5% while speed remained constant until the participant voluntarily terminated the test due to exhaustion. Each participant's VO2max was defined as the highest 30 second average value collected during the test. Heart rate at 65% of VO2max was then determined and used for the experimental trials.

Experimental procedure Participants were asked to return to the lab no earlier than 72 hours after the completion of the VO2max test to complete the first of two trials in the experimental procedure. In the 48 hours prior to each trial, participants were asked to record what they were eating, drinking and if they took any medications. All participants were asked to refrain from consuming alcohol within the 48 hours prior to the trials. With the exception of the experimental beverage, each of the two trials were identical in procedure and were separated by at least 72 hours. Testing was performed at the same time of day for each participant and all testing was completed between 4:00 and 8:00 p.m.

Participants were provided with a randomly assigned beverage containing either BCAAs or a placebo solution. Participants consumed the experimental beverage five minutes prior to their running trial. Each participant was then fitted with a HR monitor and blood was drawn three minutes after ingestion. The blood draw was immediately followed by a warm-up on the treadmill at a self-selected speed for two to five minutes. Each participant then started their 60-minute running trial at 0% incline at 65% of their established VO2max. Halfway into the 60-minute trial, each participant ingested another serving of the assigned placebo or BCAA beverage. Heart rate and the rate of perceived exertion (RPE) were collected every 10 minutes during the 60-minute trial. At the conclusion of the 60 minutes, participants cooled down for two minutes before exiting the treadmill and completing the post-exercise blood draw. Blood samples were allowed to clot for 15 minutes followed by centrifugation at 1200 RPM for 15 minutes at 4°C. The serum supernatant was then collected in clean vials and immediately stored at -80°C until liquid chromatography mass spectrometry (LCMS) analysis. Treadmill speed during the first trial were recorded and replicated during the second trial.

Experimental beverages Each participant was provided a BCAA supplement solution or a placebo solution in a double-blind, randomized crossover design. The BCAA solution was 8 oz of water mixed with approximately 8 grams of a standard BCAA supplement in powder form. Each 8-gram dose contained 2.5 grams of leucine, 1.25 grams of isoleucine and 1.25 grams of valine. The presence of BCAA was confirmed by LCMS. The placebo solution was 8 oz of water mixed with approximately 2.0 mL of a sucralose-based drink mix. Both the BCAA solution and the placebo solution were similar in color and in taste. Participants were allowed to drink additional, plain water during the 60-minute running trial if desired.

Metabolite extraction Serum samples were thawed and 20μL of serum was removed and placed in a clean vial. Protein precipitation was completed with the addition of 80μL of cold acetone followed by agitation on a vortex machine and two hours in a -80°C freezer. Serum was then centrifuged at 20,000g for 10 minutes at -4°C. The metabolite rich supernatant was collected and concentrated using negative pressure to dryness (ConcentratorPlus, Eppendorf, Hamburg, Germany). Samples were then stored at -80°C for no more than 24 hours until ready for LCMS analysis. Directly before LCMS analysis, metabolite samples were reconstituted with 40μL of methanol:water (50:50) and placed in a clean mass spectrometry vial.

LCMS conditions LCMS analysis was performed on an Agilent 6538 Q-TOF MS (Agilent Technologies, Santa Clara, CA) coupled to an Agilent 1290 UHPLC (Agilent Technologies, Santa Clara, CA) using a 1.8μm, 2.1mm X 150mm Waters HSST-3 UPLC column (Waters Corp., Milford, MA). Electrospray ionization was in positive mode. LC mobile phases were water (A), and acetonitrile (B), both with 0.1% formic acid. Flow was kept constant at 300µL per minute. The mobile phase gradient began with 95% A and finished with 5% A after seven minutes before returning to 95% at eight minutes and continuing to the end of the ten-minute run time. Column compartment temperature was kept constant at 30°C. MSMS analysis was completed using identical conditions with pooled extracted serum samples.

Data analysis Serotonin standards (Thermo Fisher Scientific, Waltham, MA) were analyzed under the described LCMS conditions and the retention time and m/z value were determined. Concentrations of 0.001µM, 0.01µM, 0.05µM, 0.1µM, 0.5µM, 1µM and 5µM were analyzed allowing for the creation of a standard concentration curve and the determination of the limit of detection. Peaks for serotonin from participant serum samples were then integrated and the concentration was calculated from the standard curve using MassHunter (Agilent Technologies, Santa Clara, CA). For the untargeted data analysis, the raw data files were converted to .mzML and .mgf files using MSConvert and then mined using mzMine. Blank samples were also created using the same metabolite procedure without serum and were analyzed under identical LCMS condition concurrently. The resulting sample blank data was also converted and mined with the sample data and were used to remove machine background and mobile phase contributions to the data. Cleaned datasets and MSMS data were then statistically analyzed using MetaboAnalyst and Sirius software, respectively. The BCAA supplement was also examined using LCMS and the results were analyzed to confirm the presence of BCAAs and additives including flavoring and sweetening agents.

Statistical Analysis Serotonin concentrations were normalized and center scaled using the caret R package. After normalization, a nested ANOVA was completed with serotonin concentration as the dependent variable and treatment and time as independent variables. The results of the nested ANOVA analysis led to further exploration of the groups and t-tests were performed between treatment and temporal groupings.

ELIGIBILITY:
Inclusion Criteria:

* Participate in at least 5 hours of cardiovascular activity per week

Exclusion Criteria:

* Any underlying injury
* The consumption of any selective serotonin re-uptake inhibitor (SSRI) medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Serotonin | 60 minutes
  Serum serotonin concentration
Untargeted metabolomics | 60 minutes
  Liquid chromatography mass spectrometry (LCMS) analysis of serum metabolites

SECONDARY OUTCOMES:
Rating of perceived exertion Borg Scale | 60 minutes
  Subjective rating of perceived exertion collected at 10 minute. Scale with values of 6-20 with intervals of 1. Low numbers indicating light exertion, high numbers indicating maximal exertion.

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Miles, PhD, Principal Investigator — Montana State University
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No